CLINICAL TRIAL: NCT05076799
Title: Effect of Lactulose and/ or Polyethylene Glycol Solution for Bowel Preparation in Colonscopy: a Multi-center Prospective Randomized Study
Brief Title: Effect of Lactulose and/or Polyethylene Glycol Solution for Bowel Preparation for Colonscopy Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan University (Other)
Collaborators: Affiliated Hospital of Southwest Medical University (Other); Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Principal Investigator, Lin Cai, Principal Investigator, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Sichuan U
Record Dates: First submitted 2021-09-03; First posted 2021-10-13 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Colonoscopy
Keywords: Polyethylene Glycols; Colonoscopy; Laxatives; Lactulose
MeSH Terms: interventions — Lactulose; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3 L Polyethylene glycol solution group (Active Comparator): The participants were instructed to consume 3000 mL of PEG solution
  Interventions: Drug: 3 L Polyethylene glycol solution
- 100 ml lactulose combined with 1 L PEG group (Experimental): the participants were instructed to consume 100 ml lactulose combined with 1000 mL of PEG solution
  Interventions: Drug: 100 ml lactulose combined with 1 L PEG
- 100 ml lactulose combined with 2 L PEG group (Experimental): the participants were instructed to consume 100 ml lactulose combined with 2000 mL of PEG solution
  Interventions: Drug: 100 ml lactulose combined with 2 L PEG
- 200 ml lactulose group (Experimental): the participants were instructed to consume 200 ml lactulose
  Interventions: Drug: 200 ml lactulose

INTERVENTIONS:
Drug: 100 ml lactulose combined with 1 L PEG — the participants were instructed to consume 100 ml lactulose combined with 1000 mL of PEG solution
  Other Names: lactulose and 1 L PEG group
  Arms: 100 ml lactulose combined with 1 L PEG group
Drug: 100 ml lactulose combined with 2 L PEG — the participants were instructed to consume 100 ml lactulose combined with 2000 mL of PEG solution
  Other Names: lactulose and 2 L PEG group
  Arms: 100 ml lactulose combined with 2 L PEG group
Drug: 200 ml lactulose — the participants were instructed to consume 200 ml lactulose alone
  Other Names: lactulose group
  Arms: 200 ml lactulose group
Drug: 3 L Polyethylene glycol solution — the participants were instructed to consume 3000 mL of PEG solution
  Other Names: control group; PEG group
  Arms: 3 L Polyethylene glycol solution group

SUMMARY:
Colonoscopy is the most useful exam used to evaluate colorectal diseases, like colorectal polyps and cancer. The appropriate bowel preparation is indispensable for colonoscopy procedures. Polyethylene glycol solution (PEG) is the most frequent laxative medication. However, the taste is poor, and patients need to drink a lot of liquids to obtain adequate visualization of the mucosal surface. In fact, no laxative has all the characteristics of an ideal medication. Lactulose is an osmotic laxative which widely used in cirrhosis and constipation patients, and could inhibit bacterial in the colon to increase colon cleanliness and prolong the effect time of PEG. Previous study demonstrate PEG combined with lactulose has a significant improvement in the quality of bowel preparation compared with PEG alone. The present study aim to assess the efficacy of lactulose with or without PEG in bowel preparation to improve mucosal visualization, reduced volume of fluid consumed, and preparation intolerance.

DETAILED DESCRIPTION:
This study will conduct in 5 clinical central. 1000 participants who were scheduled for colonoscopy age between 18 and 80 years were enrolled in the study. Exclusion criteria were patients with uncontrolled acute or recurrent chronic intestinal infections, with active gastrointestinal bleeding or gastrointestinal stricture or intestinal obstruction, with severity coronary heart disease or heart failure or renal failure and liver failure or severe electrolyte metabolism disorder, with pregnant or lactating or metal diseases or refuse to colonoscopy examination. Central stratification and block randomization is achieved via a computer-generated random-sequence table by using R software. The participants will be assigned into one of four groups at a ratio of 1 : 1, and received a single 3 L dose of either PEG or 200ml dose of lactulose, 100ml lactulose combined with 1L PEG, 100ml lactulose combined with 2L PEG. The following parameters were then obtained: time of the first defecation, defecation frequency, the overall drink liquid volume, the taste of the preparation, the tolerance evaluation, the cleansing quality of the bowel preparations and adverse reaction.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were scheduled for colonoscopy age between 18 and 80 years

Exclusion Criteria:

* uncontrolled acute or recurrent chronic intestinal infections
* active gastrointestinal bleeding, gastrointestinal stricture, intestinal obstruction
* severe electrolyte metabolism disorder, severe coronary heart disease, heart failure, renal failure or liver failure
* pregnant, lactating, have metal diseases or refuse to colonoscopy examination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The quality of bowel preparation | up to 12 months
  to assess the quality of bowel preparation by using Boston Bowel Preparation Scale. The minimum score value is 0，and the maximum value is 9. A higher score means a better outcome. Bowel cleansing was scored by the endoscopist performing the colonoscopy in the single-blind method.
The preparation intolerance | up to 12 months
  to assess the preparation intolerance including the palatability of the bowel-cleansing agents, the general satisfaction with the bowel preparation, the willingness to perform another colonoscopy by using case report questionnaire. Moreover, the ratio of drink all preparation fluids and the specific amount of bowel preparation fluid are documented.

SECONDARY OUTCOMES:
The colorectal diseases detection rate | up to 12 months
  the cecal intubation time, colonoscopy perform time, and polyp detection rate or colorectal cancer detection rate are recorded.
The adverse events | up to 12 months
  the adverse events including nausea, vomiting, abdominal pain, abdominal distension, and other adverse reactions after administration are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: juan liao, PhD, Study Director — West China Forth Hospital
Locations (1):
- west china fourth hospital of Sichuan university, Chengdu, Sichuan, China